CLINICAL TRIAL: NCT02371811
Title: Use of v Care in Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, dr mohammed elsafty, consultant, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: m2491
Record Dates: First submitted 2015-02-17; First posted 2015-02-26 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- v care group (Experimental): In this group we will use (v care) uterine manipulator during abdominal hysterectomy.
  Interventions: Device: uterine manipulator (v care)
- control group (No Intervention): In this group we will do abdominal hysterectomy without v care.

INTERVENTIONS:
Device: uterine manipulator (v care)
  Other Names: v care
  Arms: v care group

SUMMARY:
The investigators use v care during abdominal hysterectomy and evaluate its effect on duration of operation time, surgical complications and vaginal length.

ELIGIBILITY:
Inclusion Criteria:

* benign causes for hysterectomy

Exclusion Criteria:

* malignant causes for hysterectomy

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Vaginal length | within 1 week postoperative

SECONDARY OUTCOMES:
Bladder injury | within 1 week postoperative

CONTACTS AND LOCATIONS:
Overall Officials: mohammed elsafty, md, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt